CLINICAL TRIAL: NCT07401862
Title: A Phase 1, Multicenter, Open-Label, Parallel-Design Study to Assess the Pharmacokinetics and Tolerability of a Single Subcutaneous Dose of Eloralintide (LY3841136) in Participants With Mild, Moderate, or Severe Hepatic Impairment and Participants With Normal Hepatic Function
Brief Title: A Study of Eloralintide (LY3841136) in Participants With Different Levels of Liver Damage and in Participants With Healthy Livers.
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 27751; J3R-MC-YDAH (Other: Eli Lilly and Company); 2025-523847-36-00 (EU CTIS Number)
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Hepatic Insufficiency
MeSH Terms: conditions — Hepatic Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Eloralintide (Normal Hepatic Function) (Experimental): Eloralintide administered subcutaneously (SC)
  Interventions: Drug: LY3841136
- Eloralintide (Mild Hepatic Impairment) (Experimental): Eloralintide administered SC
  Interventions: Drug: LY3841136
- Eloralintide (Moderate Hepatic Impairment) (Experimental): Eloralintide administered SC
  Interventions: Drug: LY3841136
- Eloralintide (Severe Hepatic Impairment) (Experimental): Eloralintide administered SC
  Interventions: Drug: LY3841136

INTERVENTIONS:
Drug: LY3841136 — Administered SC
  Other Names: Eloralintide

SUMMARY:
The main purpose of this study is to evaluate how a medicine, LY3841136, works in participants with different levels of liver damage and in participants with healthy liver. The researchers want to see how the medicine is absorbed and used by the body, and if it causes any side effects, in participants with mild, moderate, or severe liver damage, as well as in participants with normal liver function.

For each participant, the study will last about 14 weeks, which will include a stay at the clinical research unit for 5 nights.

ELIGIBILITY:
Inclusion Criteria:

* Have a body weight of 55 kilograms (kg) or more and body mass index between 19.0 and 40.0 kilograms per square meter (kg/m²), inclusive

Group 1

* Are healthy as determined by medical history, physical examination, and other screening procedures, with clinically normal hepatic function at screening

Groups 2 through 4

* Have hepatic impairment classified as Child-Pugh score A, B, or C (mild, moderate, or severe impairment who are considered acceptable for participation in this study by the investigator. Participants must have a diagnosis of chronic hepatic impairment of greater than 6 months per physician diagnosis and standard-of-care practice, with no clinically significant changes in the opinion of the investigator within 15 days prior to screening

Participants with hepatic impairment may have stable baseline medical conditions for which neither the condition nor treatments received would negatively impact the health of the participant or study conduct

Exclusion Criteria:

* Have a history or presence of chronic or acute pancreatitis or elevation in serum amylase or lipase greater than 1.5 × upper limit of normal (ULN)
* Are pregnant or intend to become pregnant or to breastfeed during the study

Group 1

* Have liver disease, obvious clinical signs or symptoms of liver disease, acute or chronic hepatitis, or have elevations in aspartate aminotransferase (AST) or alanine transaminase (ALT) greater than 1.5 × ULN or total bilirubin (TBL) greater than 1.5 × ULN at screening
* Have a current infection with hepatitis B virus (HBV), that is,

  * if hepatitis B surface antigen (HBsAg) is positive, the participant is excluded, or
  * if HBsAg is negative and anti-Hepatitis B core antibody (HBc) is positive, further testing for HBV deoxyribonucleic acid (DNA) is required, and

    * if the screening HBV DNA is positive, the participant is excluded
* Have a current infection with hepatitis C virus (HCV), that is,

  * if anti-HCV is positive, a test for circulating HCV ribonucleic acid (RNA) is required, and
  * if HCV RNA test is positive, the participant is excluded

Groups 2, 3, and 4

* Have presence of active portal shunt or transjugular intrahepatic portosystemic shunt
* Require paracentesis more often than 2 times per month or are expected to require paracentesis during the study
* Have evidence of spontaneous bacterial peritonitis within 6 months of screening
* Have had variceal bleeding within 3 months of screening. If the participant has undergone a successful banding procedure, they may participate in the study providing at least 1 month has passed after the banding procedure at the time of screening
* Show presence of hepatocellular carcinoma
* Have hepatic encephalopathy of Grade 2 or higher
* Have TBL greater than 15 milligrams per deciliter (mg/dL)
* Have ALT greater than or equal to 6 × ULN

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Zero to Infinity AUC(0-∞) of LY3841136 | Predose on Day 1 up to Day 71
PK: Maximum Observed Drug Concentration (Cmax) of LY3841136 | Predose on Day 1 up to Day 71

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (2):
  - Orlando Clinical Research Center, Orlando, Florida
  - American Research Corporation, San Antonio, Texas
- CRU Early Phase Unit, Kistarcsa, Hungary

IPD SHARING:
Plan to Share IPD: No